CLINICAL TRIAL: NCT04957940
Title: Fish-Oil-Based Lipid Emulsion Infusion (FOBLE): Could Early Use Provide a Potential Therapy to Stop Moderate Cases of COVID-19 Diseased Patient's Shift to ICU?
Brief Title: Lipid Emulsion Infusion and COVID-19 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300631
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — SMOFlipid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMOF lipid 20% IV infusion (Experimental): Intravenous fish-oil-based lipid (SMOF lipid 20%) emulsion supplementation to standard enteral nutrition.
  Interventions: Drug: SMOFlipid
- Saline placebo IV infusion (Placebo Comparator): Intravenous 0.9% saline supplementation to standard enteral nutrition.
  Interventions: Other: 0.9% saline

INTERVENTIONS:
Drug: SMOFlipid — Intravenous fish-oil-based lipid (SMOF lipid 20%) (Fresenius Kabi, Bad Homburg, Germany) emulsion supplementation to standard enteral nutrition in a dose of 100 ml/day at a rate of 12.5 ml/h over 8 h daily for 5 days.
  Arms: SMOF lipid 20% IV infusion
Other: 0.9% saline — Receive standard enteral nutrition plus 100 ml/day 0.9% normal saline at a rate 12.5 ml/h over 8 h for 5 days
  Other Names: Normal saline
  Arms: Saline placebo IV infusion

SUMMARY:
Investigators suggest that early administration of intravenous lipid emulsion (ILE) affect the inflammatory response and improve outcome in COVID-19. The aim of this trial is to study the effect of fish-oil-based intravenous lipid emulsion (FOBLE) supplementation added to enteral nutrition on shift to ICU for upgrading oxygenation &/or ventilation in moderate cases of Covid-19 diseased patients requiring only supplemental oxygen in form of simple nasal cannula or venturi mask oxygen (during 7 days admission).

DETAILED DESCRIPTION:
A written informed consent will be taken from the patients or their relatives. Patients will be randomly assigned to receive standard enteral nutrition plus 100 ml/day 0.9% normal saline at a rate 12.5 ml/h over 8 h for 5 days as the control group (Group C) or intravenous fish-oil-based lipid (SMOF lipid 20% which contains a unique 4-oil mix containing Soya bean, Medium-chain triglycerides, Olive oil and Fish oil) (Fresenius Kabi, Bad Homburg, Germany) emulsion supplementation to standard enteral nutrition (group L) in a dose of 100 ml/day at a rate of 12.5 ml/h over 8 h daily for 5 days.Finally, 20 mL of 0.9% normal saline was injected into the burette to flush the system. The entire apparatus was disposed of when each infusion was completed. The whole process was repeated for each infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients are with diagnosis of moderate cases of covid-19 (a person who may have lower respiratory illness, such as pneumonia. However, their blood oxygen levels remain ≥94%)
* Requiring only supplemental oxygen in form of simple nasal cannula or venturi mask oxygen admitted in the intermediate care attached to our ICU with good enteral nutrition.

Exclusion Criteria:

* Hypersensitivity (peanut,eggs and soya bean)
* Uncontrolled hyperlipidemia
* Severe primary blood coagulation diseases
* Acute pancreatitis
* Acute thromboembolic diseases
* Liver failure (bilirubin >40 mmol/l, alanine aminotransferase >100 U/l and aspartate aminotransferase >100 U/l)
* RIFLE (Risk, Injury, Failure, Loss of kidney function and End-stage kidney disease) stage III and IV renal failure
* Pregnancy or lactation
* Severe neutropenia (<500 cells/mm3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-26 (Actual)

PRIMARY OUTCOMES:
Shift of patients to ICU | 7 days
  Patients will be shifted to ICU for upgrading oxygenation &/or ventilation due to failed management in the intermediate care attached to our ICU (simple nasal cannula or venturi mask oxygen).According to the Chinese diagnosis and treatment guideline for COVID-19 (trial version 7.0), severe cases were defined as including one of the following criteria: (1) respiratory frequency >30/min, (2) oxygen saturation ≤93%, and (3) PO2/FiO2 ≤300 (taking consideration that severe ARDS PO2/FiO2 ratio < 100). Severe patients who need higher levels of oxygen support (high-flow nasal cannula HFNC or non invasive continuous positive airway pressure CPAP) to correct hypoxemia, or multiple organ dysfunction, are admitted to the ICU.

SECONDARY OUTCOMES:
Percentage of short-term outcome | 7 days
  Assessing the percentage % of short-term outcome for cases admitted in the intermediate care attached to our ICU and numbers of patients either died, shifted to ICU for upgrading oxygenation and or ventilation or discharged to home.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, MD, Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Simopoulos AP. Omega-3 fatty acids in inflammation and autoimmune diseases. J Am Coll Nutr. 2002 Dec;21(6):495-505. doi: 10.1080/07315724.2002.10719248. PMID 12480795